CLINICAL TRIAL: NCT00756184
Title: 1-year Randomized Control Trial Investigating the Value of an Intervention to Enhance Adherence in Glaucoma Patients Receiving Prostaglandin Monotherapy and in Patients Who Are Candidates for Adjunctive Therapy
Brief Title: Value of an Intervention to Enhance Adherence in Glaucoma Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A5133
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Glaucoma
Keywords: Glaucoma; Adherence; Teaching
MeSH Terms: conditions — Glaucoma | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Intervention will consist of intensive teaching on the nature of glaucoma, value of IOP control, need to adhere to medical therapy and counseling on the proper use of travoprost eye drops.
  Interventions: Device: TDA adherence monitor for travoprost therapy
- B (Placebo Comparator): Intervention with travoprost therapy and TDA monitoring. Patients of this arm will also be prescribed travoprost and will be followed up in a standard clinical fashion. This group will receive a comparable amount of personal physician attention, but will not be given adherence, or glaucoma education and will not be told that their adherence will be monitored. Their attention placebo intervention will discuss the importance and techniques of good "eye health" (sunglasses, vitamins, cataract development, etc but no details, or discussion of either glaucoma or adherence) will insure that the study results are not a result of a change in physician attention to a patient, per se, rather than adherence training.
  Interventions: Device: TDA and travoprost monotherapy

INTERVENTIONS:
Device: TDA adherence monitor for travoprost therapy — monitoring adherence to travoprost therapy
  Other Names: Adherence and IOP control after 12 months of therapy
  Arms: A
Device: TDA and travoprost monotherapy — Patients will be prescribed travoprost therapy and will be followed up in a standard clinical fashion with a attention placebo at both baseline and 6 months
  Arms: B

SUMMARY:
A one-year, randomized, attention placebo-controlled trial investigating the value of comprehensive adherence specific interventions, over the course of one year, to enhance adherence in both (a) newly diagnosed open-angle glaucoma, or ocular hypertension patients, naive to medical therapy and (b) those who have failed monotherapy with any prostaglandin analogue (and are therefore candidates for adjunctive therapy) who then are randomized to receive only travoprost monotherapy. Subjects will be randomized to two different interventions involving direct physician education, each of which will take approximately the same amount of physician time: The first will be intensive adherence education that will continue throughout the year. The second will be intensive eye care education, but without any direct adherence education. All patients participating in the study will be monitored for adherence by the TDA. The study will demonstrate for the first time the role of adherence-specific training in improving patient adherence and will validate the TDA in monitoring and improving adherence in glaucoma. This will correlate with prior work that has documented that greater adherence is associated with marked improvement in intraocular pressure (IOP) control. A second goal will be seeing whether improving adherence will change the course of glaucoma therapy by making therapeutic failures into therapeutic successes by reducing the need for adjunctive therapy using only monotherapy with travoprost.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with glaucoma
* Suboptimally controlled patients with glaucoma
* Untreated baseline IOP greater than 21 mm Hg but less than 32 mm Hg
* Patients who have not responded satisfactorily to PGA therapy
* Patients who are about to have adjunctive therapy administered
* Patients who consent to participate in this trial

Exclusion Criteria:

* Glaucoma patients with high pressure
* Advanced glaucoma
* Patients with side effects to PGA therapy
* Unwilling to participate

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-09; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Adherence rate between intervention and control groups | 1,3,6,12 months

SECONDARY OUTCOMES:
IOP control | 12 months
  Monitoring of morning IOP control between the active and the control groups

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios G Konstas, MD, PhD, Principal Investigator — Glaucoma Unit, 1st University Dept AUT